CLINICAL TRIAL: NCT02615639
Title: A Clinical Trial on Hepatitis B Vaccine Activated-Dendritic Cells Combined With Anti-HBV Drugs in Chronic Hepatitis B
Brief Title: A Clinical Trial on Hepatitis B Vaccine Activated-Dendritic Cells Combined With Anti-HBV Drugs in CHB
Acronym: CTHBVACADCHB
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yuehua Huang, chief director of liver Lab, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SunYatSenIDD
Record Dates: First submitted 2015-11-12; First posted 2015-11-26 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Hepatitis B
Keywords: HPDC-T cells; CHB; immuno therapy
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; peginterferon alfa-2a; Telbivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- HPDC-T cells & entecavir (Experimental): HPDC-T cells 1-5×10^5 intravenous injection, every 2 weeks for 24 weeks , and entecavir(ETV) 0.5mg tablet by mouth, every night.
  Interventions: Biological: HPDC-T cells & Entecavir
- entecavir (Active Comparator): entecavir 0.5mg tablet by mouth, every night.
  Interventions: Drug: Entecavir
- HPDC-T cells & IFN-a-2a (Experimental): HPDC-T cells 1-5×10^5 intravenous injection, every 2 weeks for 24 weeks ,and IFN-a-2a 180ug subcutaneous injection， every week for 9 months.
  Interventions: Drug: HPDC-T cells & IFN-a-2a
- IFN-a-2a (Active Comparator): IFN-a-2a 180ug subcutaneous injection， every week for 9 months.
  Interventions: Drug: IFN-a-2a
- HPDC-T cells & Telbivudine (Experimental): HPDC-T cells 1-5×10^5 intravenous injection, every 2 weeks for 24 weeks ,and Telbivudine 600mg tablet by mouth, every night.
  Interventions: Drug: HPDC-T cells & Telbivudine
- Telbivudine (Active Comparator): Telbivudine 600mg tablet by mouth, every night.
  Interventions: Drug: Telbivudine

INTERVENTIONS:
Biological: HPDC-T cells & Entecavir — experimental groups will be given HPDC-T cells & Entecavir. HPDC-T cells will be given for 24weeks on the basis of anti-HBV therapy ,and entecavir 0.5mg tablet every night by mouth
  Other Names: Hepatitis B Vaccine Activated-DCs & Entecavir
  Arms: HPDC-T cells & entecavir
Drug: Entecavir — 0.5mg tablet every night by mouth
  Other Names: Baraclude
  Arms: entecavir
Drug: HPDC-T cells & IFN-a-2a — experimental groups will be given HPDC-T cells & IFN-a-2a. HPDC-T cells will be given for 24 weeks on the basis of anti-HBV therapy ,and IFN-a-2a 180ug subcutaneous injection every week
  Other Names: Hepatitis B Vaccine Activated-DCs & Pegasys
  Arms: HPDC-T cells & IFN-a-2a
Drug: IFN-a-2a — IFN-a-2a 180ug subcutaneous injection every week
  Other Names: Pegasys
  Arms: IFN-a-2a
Drug: HPDC-T cells & Telbivudine — experimental groups will be given HPDC-T cells & Telbivudine. HPDC-T cells will be given for 24weeks on the basis of anti-HBV therapy ,and Telbivudine 600mg tablet every day by mouth
  Other Names: Hepatitis B Vaccine Activated-DCs & Telbivudine
  Arms: HPDC-T cells & Telbivudine
Drug: Telbivudine — Telbivudine 600mg tablet every day by mouth
  Other Names: LDT
  Arms: Telbivudine

SUMMARY:
The anti-virus effects is not satisfying in some of Chronic Hepatitis B（CHB) patients who have been on anti-Hepatitis B Virus (HBV) drugs therapy. Dendritic cell (DC) is critical in Hepatitis B Virus (HBV) specific immunity in the process of producing HBV promoter specific cytotoxic T cells (CTLs) and specific T helper cells (HTLs), however they are defective in CHB patients. Therefore, if it were going to remove HBV completely, it mainly depends if the body itself can produce enough HBV specific cytotoxic T cells (CTLs) and specific T helper cells (HTLs). Our research is to plus Hepatitis B Vaccine Activated-DCs therapy to CHB patients who have been on anti-HBV drugs but with poor effects, supposing to significantly improve anti-HBV efficacy, even to clean HBV from the patients.

DETAILED DESCRIPTION:
Patients who have been on anti-HBV therapy Complying with the inclusion criteria will be enrolled into our research, Nucleoside analogues (NAs,entecavir） treatment for more than 1 year or interferon（IFN)-a-2a (IFN-a-2a,Pegasys） treatment for more than 24 weeks. The patients will be randomly assigned to experimental group and control group with the ratio of 2:1, one group (control group) will go on receive the anti-HBV drugs treatment solely; another group (experimental group) after enrollment will immediately receive the Hepatitis B Vaccine activated-DCs (HPDC-T cells) for 24 weeks (every 2 weeks once for 24 weeks, 12 times in total), at the same time co-use anti-HBV drugs treatment, as for Pegasys, it will go on to be used for 12 weeks after HPDC-T cells treatment completed.

The technical route of HBV-T cells prepared: First, investigators collect fresh blood of CHB, mononuclear cells were isolated, and induced to HBsAg pulsed DCs in Hepatitis B vaccine (Shenzhen kangtai, Shenzhen, China) and interleukin-4（IL-4)/granulocyte-macrophage colony-stimulating factor(GM-CSF） (Perprotech, New Jersey, USA) (7 days), then co-culture of DCs and Peripheral Blood Mononuclear Cell(PBMCs ）7days, obtain HBV specific T cells, return to the patient finally.

ELIGIBILITY:
Inclusion Criteria:

* chronic hepatitis B patients, aged 18~65，Chinese
* have been on entecavir（ETV） or telbivudine（LDT） treatment for more than 1 year,and HBV DNA<100 IU/ml（Roche Cobas）;or have been on
* have been on PEG-IFN treatment for more than 24 weeks,and 20 < HBV DNA < 20000 IU/ml（Roche Cobas）.
* HBsAg 100~5000 IU/ml
* HBeAg 10~500 COI

Exclusion Criteria:

* Superinfection or co-infection with hepatitis A, C, D, E, cytomegalovirus and HIV, or Epstein-Barr virus;
* other liver diseases such as alcoholic liver disease, drug-induced hepatitis, Wilson disease and autoimmune hepatitis;
* ascites or gastrointestinal bleeding or peptic ulcer or esophageal varix by electronic gastroscope examination;
* liver cirrhosis (including compensated and decompensated cirrhosis) and liver failure;
* severe bacterial or fungal infections;
* a history of diabetes or cardiac disease or hypertension or nephrosis;
* pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Hepatitis B surface Antigen （HBeAg）seroconversion | 3 years
  to increase Hepatitis B surface antigen (HBsAg) loss rate from 1% up to 11% or more

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by low-grade fever, Infection and shock. | one and a half year
  Safety profiles include side effects of anti-HBV drugs(ETV,LDT and IFN-a), viral resistance of anti-HBV drugs. And side effects of HPDC-T cells infusion,such as low-grade fever, Infection and shock.The difference of side effects rates between anti-HBV drugs monotherapy and anti-HBV drugs plus HPDC-T cells combined therapy will also be analyzed.
Hepatitis B envelope Antigen （HBeAg） seroconversion | 3 years
  to increase HBeAg negative rate by 12 percentage points on the basis of the existing data
HBV DNA clearance | 3 years
  to increase the undetectable rate of HBV DNA
ALT recovery | 3 years
  to increase the recovery rate of ALT

CONTACTS AND LOCATIONS:
Overall Officials: Lubiao Chen, MD.&PHD., Principal Investigator — The Third Affiliated Hospital of Sun Yet-sun University

REFERENCES:
- [Background] Luo J, Li J, Chen RL, Nie L, Huang J, Liu ZW, Luo L, Yan XJ. Autologus dendritic cell vaccine for chronic hepatitis B carriers: a pilot, open label, clinical trial in human volunteers. Vaccine. 2010 Mar 16;28(13):2497-504. doi: 10.1016/j.vaccine.2010.01.038. Epub 2010 Jan 29. PMID 20117267
- [Background] Akbar SM, Furukawa S, Horiike N, Abe M, Hiasa Y, Onji M. Safety and immunogenicity of hepatitis B surface antigen-pulsed dendritic cells in patients with chronic hepatitis B. J Viral Hepat. 2011 Jun;18(6):408-14. doi: 10.1111/j.1365-2893.2010.01320.x. PMID 20487261